CLINICAL TRIAL: NCT00186095
Title: Mixed Chimeric Transplantation for Primary Amyloidosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed, never started.
Sponsor: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT129
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Amyloidosis
Keywords: Amyloidosis; nonmyeloablative; hematopoietic; cell transplantation
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: autologous followed by nonmyeloablative allogeneic transplant

SUMMARY:
To evaluate the role of nonmyeloablative allogeneic transplantation in Amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* primary amyloidosis
* adequate organ function
* matched sibling donor

Exclusion Criteria:

* evidence of multiple myeloma
* HIV positive

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2000-12; Study Completion 2006-09

PRIMARY OUTCOMES:
Treatment of patients with nonmyeloablative allogeneic transplant for amyloidosis.

SECONDARY OUTCOMES:
Toxicity of therapy
Changes in marrow and serum abnormalities
Improvement in end-organ function.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Stockerl-Goldstein, MD, Principal Investigator — Stanford University